CLINICAL TRIAL: NCT05648253
Title: Pilot Study to Assess the Feasibility of Use of a Novel Vaginal Dilator Device Post-radiation for Patients With Pelvic Malignancies
Brief Title: Feasibility of Hyivy Device Post-Radiation for Pelvic Malignancies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hyivy Health Inc (Industry)
Collaborators: Grand River Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYV-002-C23
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Vaginal Stenosis; Radiation Therapy; Cancer; Pelvic Pain; Pelvic Cancer
Keywords: Dilator; Post radiation therapy
MeSH Terms: conditions — Neoplasms; Pelvic Pain; Pelvic Neoplasms

STUDY DESIGN:
Intervention Model Description: A prospective single-arm pre/post repeated-measures pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hyivy Intravaginal Device (Experimental): Participants will receive a Hyivy intravaginal device for at-home use. Recommended use is three times per week for 12 weeks and consists of 10 minutes of heat (37-39ºC) and 10 minutes of dilation per session.
  Interventions: Device: Hyivy Intravaginal Device

INTERVENTIONS:
Device: Hyivy Intravaginal Device — Intravaginal use of Hyivy device three times per week for 12 weeks, with each session consisting of 10 minutes of heat (37-39ºC) and 10 minutes of dilation.

SUMMARY:
Vaginal dilator therapy (VDT) with static dilators is often prescribed to patients following vaginal or pelvic radiation therapy. This study seeks to evaluate the feasibility of a novel intravaginal device that delivers patient-controlled dilation (Hyivy device). The study is designed as a proof-of-concept single-arm pilot study. The primary objective is to assess safety and tolerability, while also evaluating changes in health-related quality of life and pelvic pain.

DETAILED DESCRIPTION:
Radiation therapy is a common treatment for cancer in the pelvic area and is considered a mainstay of treatment for cancers of the cervix, uterus, and anorectum. Patients with a vagina and vaginal canal who undergo vaginal or pelvic radiation therapy are at risk for developing vaginal stenosis, defined in part by a shortening and/or narrowing of the vaginal canal, which can lead to damaged tissue and pain with examination/vaginal penetration.

Vaginal dilator therapy (VDT) is prescribed to prevent vaginal stenosis. Adherence to VDT in the months following radiation is quite low. Reasons may include limited size options of static dilators, lack of time, general fatigue, emotional well-being, and associating dilator use with underlying malignancy and radiation treatment. Alternatives to static dilators that are safe and effective may improve adherence to VDT and improve patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age ≥ 18 at the time of enrollment
* 2.Patient with a vagina or vaginal canal who have completed radiation therapy (either external beam or brachytherapy, or a combination of both) for endometrial cancer, cervical cancer, anal cancer, or rectal cancer, without concomitant chemotherapy
* 3.Generally in good health (other than due to cancer), at the discretion of the investigator(s)
* 4.Eastern Cooperative Oncology Group (ECOG) score or 0 to 2
* 5.Participants must be post-menopausal (natural or surgically) for at least 1 year prior to screening or be surgically sterile (absence of ovaries and/or uterus); or, a participant of child-bearing potential must agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months.
* 6.Agree not to use other dilators for the 12-week intervention period
* 7.Must have the ability to charge the investigational device
* 8.Must be willing and able to insert intravaginal device
* 9.Able to understand, comply and consent to protocol requirements and instructions
* 10.Able to attend scheduled study visits and complete required investigations
* 11.Ability to understand and willingness to sign written informed consent

Exclusion Criteria:

* 1.Participants who are pregnant or planning to become pregnant during the trial
* 2.Any major surgery in the past 3 months unless post-surgery dilator use is recommended by a physician, or anticipates having a major surgery during the study
* 3.Any other medical condition or clinical finding giving reasonable suspicion of a disease or condition that contraindicates the use of the investigational product or that may affect the interpretation of the results or leave the patient at high risk from treatment complications, at the discretion of the investigator(s)
* 4.Allergy to Hyivy device's materials
* 5.Active pelvic or gynaecological infection
* 6.Current use of antibiotics for any infection
* 7.Have open wounds, cuts, or open sores present in the vaginal or pelvic area
* 8.Severe atrophic vaginitis or very dry, itchy, or sore vagina/vaginal area, at the discretion of the investigator(s)
* 9.Hypoesthesia or loss in sensation of the pelvic floor
* 10.Total and/or partial prolapse of the uterus and/or vagina
* 11.Symptoms of severe urinary retention, severe extra-urethral incontinence, or overflow incontinence
* 12.Unable to position the device according to directions for use
* 13.Use of any medical devices that may interfere with the investigational device's function, such as pacemakers, ventilators, and ear implants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 12 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of the Hyivy device | Up to 12-weeks
  Occurrence of adverse events (AE) and serious adverse events (SAE).

SECONDARY OUTCOMES:
Quality of Life (FACT-G) | Baseline, 6-weeks, 12-weeks
  Changes in health-related quality of life (HRQoL) as assessed by the Functional Assessment of Cancer Therapy - General (FACT-G).
Pelvic pain (VAS) | Baseline, 6-weeks, 12-weeks
  Changes in pelvic pain as assessed by a visual analog scale (VAS).
Adherence to study protocol | 6-weeks, 12-weeks
  Usage data collected by the Hyivy device will be used to assess participant adherence to the study regimen of 3 times/week device use.

OTHER OUTCOMES:
Device usability and patient satisfaction | 12-weeks
  Study-specific questionnaire to gather patient feedback

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Glick, MD, Principal Investigator — Grand River Hospital
Locations (1):
- Grand River Regional Cancer Centre, Waterloo Regional Health Network @ Midtown, Kitchener, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers

REFERENCES:
- [Background] Damast S, Jeffery DD, Son CH, Hasan Y, Carter J, Lindau ST, Jhingran A. Literature Review of Vaginal Stenosis and Dilator Use in Radiation Oncology. Pract Radiat Oncol. 2019 Nov;9(6):479-491. doi: 10.1016/j.prro.2019.07.001. Epub 2019 Jul 11. PMID 31302301
- [Background] International Clinical Guideline Group. International Guidelines on Vaginal Dilation after Pelvic Radiotherapy.; 2012. https://owenmumford.com/us/wp-content/uploads/sites/3/2014/11/Dilator-Best-Practice-Guidelines.pdf.
- [Background] Law E, Kelvin JF, Thom B, Riedel E, Tom A, Carter J, Alektiar KM, Goodman KA. Prospective study of vaginal dilator use adherence and efficacy following radiotherapy. Radiother Oncol. 2015 Jul;116(1):149-55. doi: 10.1016/j.radonc.2015.06.018. Epub 2015 Jul 8. PMID 26164775
- [Background] Bakker RM, Vermeer WM, Creutzberg CL, Mens JW, Nout RA, Ter Kuile MM. Qualitative accounts of patients' determinants of vaginal dilator use after pelvic radiotherapy. J Sex Med. 2015 Mar;12(3):764-73. doi: 10.1111/jsm.12776. Epub 2014 Nov 25. PMID 25424559
- [Background] Araya-Castro P, Sacomori C, Diaz-Guerrero P, Gayan P, Roman D, Sperandio FF. Vaginal Dilator and Pelvic Floor Exercises for Vaginal Stenosis, Sexual Health and Quality of Life among Cervical Cancer Patients Treated with Radiation: Clinical Report. J Sex Marital Ther. 2020;46(6):513-527. doi: 10.1080/0092623X.2020.1760981. Epub 2020 May 2. PMID 32364016